CLINICAL TRIAL: NCT05257096
Title: Can Medical Clowns Prevent the Usage of Sedation During the Performance of EEG in Young Children
Brief Title: Performance of EEG in Children With Medical Clowns
Acronym: MECLEES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Director Pediatric Departement, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: bnz 049-19
Record Dates: First submitted 2022-01-30; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: EEG With Periodic Abnormalities; Child, Only
Keywords: EEG with Periodic Abnormalities; Play Role; Child, Only

STUDY DESIGN:
Intervention Model Description: The children will be divided to either group randomly according to the day of the test.
  1. 50 Children performing the EEG at the days that the medical clown is available will be included in the study group.
  2. 50 Children performing the EEG at the days that the medical clown is unavailable will be included in the control group.
Who Masked: Investigator
Masking Description: The EEG reading will be blinded to the intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical clown EEG (Experimental): 50 Children performing the EEG at the days that the medical clown is available will be included in the study group.
  Interventions: Behavioral: Medical clown
- Regular EEG (No Intervention): 50 Children performing the EEG at the days that the medical clown is unavailable will be included in the control group. The EEG will be performed in the traditional way without medical clowns.

INTERVENTIONS:
Behavioral: Medical clown — The medical clown will meet the children in the waiting room for 15-30 minutes and will accompany them through the whole investigation, up to one hour.
  Other Names: non
  Arms: Medical clown EEG

SUMMARY:
EEG is an important test in the diagnosis epilepsy. The test does not hart, however many electrodes are attached to the child's scalp and situation is stressful. In order to achieve cooperation some use sedative drugs such as Chloralhydrate in young children. The investigetors believe that the integration of medical clowns in the EEG test can distract the children from the stressful environment and encourage them to cooperate. This can prevent the need of using sedation, can improve the quality of the test and improve the child's and parent's experience. One hundred children ages 1-10 years of age performing EEG test at the Bnai Zion medical center will be randomly divided into two groups. One group will the perform the test in the regular practice, and in the other half, medical clowns will be part of the test. The process will be rated by the child, his parents, the EEG technician and the physician reading the EEG. The two groups will be compared in all assessed measures through a statistical analysis.

DETAILED DESCRIPTION:
Can Medical Clowns prevent the usage of sedation during the performance of EEG in Young Children MECLEES - MEdical CLowns EEg Study

The study will be performed at the Pediatric Neurology Unit in Bnai Zion Medical Center, Haifa, Israel.

Purpose The aim our study is to investigate the performance of EEG in young children in cooperation with medical clowns. Can the presence of a medical clown prevent the need of using sedation? Does it improve the child's and parent's experience? Does it improve the quality of the test?

Study procedure The children will be divided to either group randomly according to the day of the test.

1. 50 Children performing the EEG at the days that the medical clown is available will be included in the study group.
2. 50 Children performing the EEG at the days that the medical clown is unavailable will be included in the control group.

Study group: The medical clown will meet the children in the waiting room for 15-30 minutes and will accompany them through the whole investigation, up to one hour.

Control group: children that will perform EEG without a medical clown, will perform it either with sedation or without one according to the common practice.

Outcome measures

The following parameters will be assessed (Appendix 1-4):

1. Child anxiety using mYPAS (10-11) for assessing child anxiety questionnaire.
2. Parent's satisfaction.
3. Technician's evaluation.
4. EEG quality will be evaluated by both technicians and the physicians independently. The physician will be blinded to the presence of a medical clown during the test.

Ethical consideration:

Prior to study ignition IRB approval will be obtained. Any change in the study protocol must be re-approved by the IRB.

All patients enrolled to the study must provide their written consent prior to entering the study. The informed consent will be signed by the parents and retained by the investigator as a part of the study records.

No records of names or identification will be published.

Statistical analysis The study will be randomized and controlled. The physician assessing the EEG will be blinded, however the child, his parents and the EEG technician's will not be blinded. Study and control groups will be compared via independent t-tests, significance will be considered if p<0.05.

ELIGIBILITY:
Inclusion Criteria

* Children age 1-10 years
* Undergoing EEG test at the Bnai Zion Medical Center.

Exclusion Criteria

* Children younger than 1 year or older than 10 years
* Children using sedation for the test.
* A child or a family that refuses to participate initially or during the test.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 2 years
  Child anxiety using the modified Yale Preoperative Anxiety Scale ( mYPAS 5-22 points, higher scores reflects anxity) for assessing child anxiety questionnaire.
EEG quality | 2 years
  Electroencephalogram (EEG) quality will be evaluated by both technicians and the physicians independently in 1-5 likert sclae (1-best 5- worst). The physician will be blinded to the presence of a medical clown during the test.

SECONDARY OUTCOMES:
Parent's satisfaction during EEG procedure | 2 Years
  Parent's satisfaction from the procedure on 1-5 likert sclae (1-best 5- worst).
Technician's satisfaction during EEG procedure | 2 Years
  Technician's satisfaction from the procedure on 1-5 likert sclae (1-best 5- worst).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob genizi, md, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bornstein Y. [Medical clowns at hospitals and their effect on hospitalized children]. Harefuah. 2008 Jan;147(1):30-2, 95, 94. Hebrew. PMID 18300620
- [Result] Britton JW, Kosa SC. The clinical value of chloral hydrate in the routine electroencephalogram. Epilepsy Res. 2010 Feb;88(2-3):215-20. doi: 10.1016/j.eplepsyres.2009.11.012. Epub 2009 Dec 23. PMID 20031374
- [Result] Olson DM, Sheehan MG, Thompson W, Hall PT, Hahn J. Sedation of children for electroencephalograms. Pediatrics. 2001 Jul;108(1):163-5. doi: 10.1542/peds.108.1.163. PMID 11433070
- [Result] Sanborn PA, Michna E, Zurakowski D, Burrows PE, Fontaine PJ, Connor L, Mason KP. Adverse cardiovascular and respiratory events during sedation of pediatric patients for imaging examinations. Radiology. 2005 Oct;237(1):288-94. doi: 10.1148/radiol.2371041415. PMID 16183936
- [Result] Malviya S, Voepel-Lewis T, Prochaska G, Tait AR. Prolonged recovery and delayed side effects of sedation for diagnostic imaging studies in children. Pediatrics. 2000 Mar;105(3):E42. doi: 10.1542/peds.105.3.e42. PMID 10699144
- [Result] Cote CJ, Notterman DA, Karl HW, Weinberg JA, McCloskey C. Adverse sedation events in pediatrics: a critical incident analysis of contributing factors. Pediatrics. 2000 Apr;105(4 Pt 1):805-14. doi: 10.1542/peds.105.4.805. PMID 10742324
- [Result] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685
- [Result] Golan G, Tighe P, Dobija N, Perel A, Keidan I. Clowns for the prevention of preoperative anxiety in children: a randomized controlled trial. Paediatr Anaesth. 2009 Mar;19(3):262-6. doi: 10.1111/j.1460-9592.2008.02903.x. Epub 2008 Dec 23. PMID 19143948
- [Result] Dvory A, Goshen Y, Ruimi S, Bikov S, Halevy R, Koren A. Dream Doctor Intervention Instead of Sedation: Performing Radionuclide Scanning Without Sedation in Young Children: A Study in 142 Patients. J Altern Complement Med. 2016 May;22(5):408-12. doi: 10.1089/acm.2015.0090. Epub 2016 Mar 30. PMID 27028874
- [Result] Wassmer E, Carter PF, Quinn E, McLean N, Welsh G, Seri S, Whitehouse WP. Melatonin is useful for recording sleep EEGs: a prospective audit of outcome. Dev Med Child Neurol. 2001 Nov;43(11):735-8. doi: 10.1017/s0012162201001347. PMID 11730146
- [Result] Loewy J, Hallan C, Friedman E, Martinez C. Sleep/sedation in children undergoing EEG testing: a comparison of chloral hydrate and music therapy. Am J Electroneurodiagnostic Technol. 2006 Dec;46(4):343-55. PMID 17285817
- [Result] Slifer KJ, Avis KT, Frutchey RA. Behavioral intervention to increase compliance with electroencephalographic procedures in children with developmental disabilities. Epilepsy Behav. 2008 Jul;13(1):189-95. doi: 10.1016/j.yebeh.2008.01.013. Epub 2008 Mar 17. PMID 18348911
- [Result] Fong CY, Lim WK, Li L, Lai NM. Chloral hydrate as a sedating agent for neurodiagnostic procedures in children. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD011786. doi: 10.1002/14651858.CD011786.pub3. PMID 34397100
- [Result] Goldberg A, Stauber T, Peleg O, Hanuka P, Eshayek L, Confino-Cohen R. Medical clowns ease anxiety and pain perceived by children undergoing allergy prick skin tests. Allergy. 2014 Oct;69(10):1372-9. doi: 10.1111/all.12463. Epub 2014 Aug 4. PMID 24943088
- [Result] Meiri N, Ankri A, Hamad-Saied M, Konopnicki M, Pillar G. The effect of medical clowning on reducing pain, crying, and anxiety in children aged 2-10 years old undergoing venous blood drawing--a randomized controlled study. Eur J Pediatr. 2016 Mar;175(3):373-9. doi: 10.1007/s00431-015-2652-z. Epub 2015 Oct 16. PMID 26475347
- [Result] Newman N, Kogan S, Stavsky M, Pintov S, Lior Y. The impact of medical clowns exposure over postoperative pain and anxiety in children and caregivers: An Israeli experience. Pediatr Rep. 2019 Sep 24;11(3):8165. doi: 10.4081/pr.2019.8165. eCollection 2019 Sep 24. PMID 31579203
- [Result] Ben-Pazi H, Cohen A, Kroyzer N, Lotem-Ophir R, Shvili Y, Winter G, Deutsch L, Pollak Y. Clown-care reduces pain in children with cerebral palsy undergoing recurrent botulinum toxin injections- A quasi-randomized controlled crossover study. PLoS One. 2017 Apr 17;12(4):e0175028. doi: 10.1371/journal.pone.0175028. eCollection 2017. PMID 28414728
- [Result] Gjaerde LK, Hybschmann J, Dybdal D, Topperzer MK, Schroder MA, Gibson JL, Ramchandani P, Ginsberg EI, Ottesen B, Frandsen TL, Sorensen JL. Play interventions for paediatric patients in hospital: a scoping review. BMJ Open. 2021 Jul 26;11(7):e051957. doi: 10.1136/bmjopen-2021-051957. PMID 34312210
- [Result] Fernandes SC, Arriaga P. The effects of clown intervention on worries and emotional responses in children undergoing surgery. J Health Psychol. 2010 Apr;15(3):405-15. doi: 10.1177/1359105309350231. PMID 20348361
- [Result] Lopes-Junior LC, Silveira DSC, Olson K, Bomfim EO, Veronez LC, Santos JC, Alonso JB, Nascimento LC, Pereira-da-Silva G, Lima RAG. Clown Intervention on Psychological Stress and Fatigue in Pediatric Patients With Cancer Undergoing Chemotherapy. Cancer Nurs. 2020 Jul/Aug;43(4):290-299. doi: 10.1097/NCC.0000000000000690. PMID 30801267
- [Result] He HG, Zhu L, Chan SW, Klainin-Yobas P, Wang W. The effectiveness of therapeutic play intervention in reducing perioperative anxiety, negative behaviors, and postoperative pain in children undergoing elective surgery: a systematic review. Pain Manag Nurs. 2015 Jun;16(3):425-39. doi: 10.1016/j.pmn.2014.08.011. PMID 26025800
- [Result] Godino-Ianez MJ, Martos-Cabrera MB, Suleiman-Martos N, Gomez-Urquiza JL, Vargas-Roman K, Membrive-Jimenez MJ, Albendin-Garcia L. Play Therapy as an Intervention in Hospitalized Children: A Systematic Review. Healthcare (Basel). 2020 Jul 29;8(3):239. doi: 10.3390/healthcare8030239. PMID 32751225
- [Result] Koukourikos K, Tzeha L, Pantelidou P, Tsaloglidou A. THE IMPORTANCE OF PLAY DURING HOSPITALIZATION OF CHILDREN. Mater Sociomed. 2015 Dec;27(6):438-41. doi: 10.5455/msm.2015.27.438-441. PMID 26889107
- [Derived] Jacob G, Einav B, Ashy M, Nofar MA, Aviad S, Ayed M. The beneficial effect of medical clowns on performance of EEG in young children: a randomized controlled study. Eur J Pediatr. 2022 Sep;181(9):3449-3457. doi: 10.1007/s00431-022-04555-z. Epub 2022 Jul 15. PMID 35838778